CLINICAL TRIAL: NCT06095661
Title: Immersive Virtual Reality to Decrease Postoperative Pain in Older Adults Following Elective Major Surgery: A Feasibility and Acceptability Study
Brief Title: Virtual Reality as a Postoperative Pain Management Adjunct in Older Adults: An Acceptability and Feasibility Study
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-39037
Record Dates: First submitted 2023-08-13; First posted 2023-10-23 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Aged; Surgery; Pain, Postoperative; Virtual Reality
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxymetholone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality (Experimental): Each enrolled participant in a single arm will be offered a virtual reality headset with a menu of virtual reality environments and experiences such as nature scenes, mindful meditation, travel, and various games. Enrolled participants be offered the virtual reality as early as the first day after their inpatient surgery in their hospital room. Each virtual reality session will last 5-30 minutes, depending on the participant's selection of the virtual reality environment/experience. Participants will have the option to use the virtual reality as often as twice daily up through the third day after their surgery during their hospitalization, for a total of six sessions.
  Interventions: Other: REAL System i-Series VR head-mounted display (HMD) from Penumbra, Inc.

INTERVENTIONS:
Other: REAL System i-Series VR head-mounted display (HMD) from Penumbra, Inc. — The VR intervention will use the REAL System i-Series VR head-mounted display (HMD) with built-in audio purchased from Penumbra, Inc. The i-Series is a gazed-controlled and fully immersive VR headset preloaded with immersive environments that promote positive distraction and relaxation through interactive experiences. These VR experiences include mindful meditation, travel, various nature scenes, and game experiences. REAL i-Series is classified as an unclassified product with product code PWC, a general wellness product FDA #3005168196.

SUMMARY:
This single-arm mixed methods study aims to determine potential differences in self-reported postoperative pain intensity levels, anxiety, and state of relaxation through immediate pre-post intervention evaluation among those aged 65 or older who receive immersive virtual reality during their hospitalization, up to three days following major elective surgery. In addition, the investigators will evaluate the feasibility and acceptability of virtual reality for use in this older adult population. This study will not evaluate the efficacy of VR.

The main questions this study seeks to answer are:

1. What is the feasibility and acceptability of using immersive virtual reality to impact clinical outcomes such as pain, anxiety, and relaxation in older adults who have undergone major elective surgery?
2. What is the older adult's user experience with virtual reality during hospitalization up to the three days following major elective surgery?

DETAILED DESCRIPTION:
Current treatment options for postoperative pain in older adults tend to be concentrated on opioid and opioid-sparing medications, which carry an increased risk of complications in older adults. One non-pharmacological intervention to manage acute pain that has recently emerged in the healthcare setting is virtual reality (VR).VR engages the user through various technological equipment with differing degrees of immersion and has demonstrated efficacy in decreasing acute pain in various clinical settings, such as burn wound care treatment and adult and pediatric medical procedures. However, there is a scarcity of research examining VR as an adjunct treatment in older adult populations. Therefore, this study aims to examine the acceptability and efficacy of VR as a possible adjunct to current postoperative pain management regimens in older surgical patients undergoing inpatient elective major operations.

The overarching hypotheses are: 1. Older adults who receive immersive VR will demonstrate immediate improvements in self-reported pain intensity, anxiety, and state of relaxation from pre-intervention levels, and 2. Older adults will consider their VR experience positive, effective, and practical in the inpatient postoperative period, with negligible side effects reported.

The VR intervention will consist of the use of the REAL System i-Series VR head-mounted display (HMD) with built-in audio purchased from Penumbra, Inc. The i-Series is a gazed-controlled and fully immersive VR headset preloaded with immersive environments that promote positive distraction and relaxation through interactive experiences. These VR experiences include mindful meditation, travel, various nature scenes, and game experiences. After written informed consent is obtained and baseline questionnaires have been completed, enrolled participants will be given the option to utilize the REAL i-series HMD during their postoperative inpatient stay on the medical-surgical unit, as early as the first day following surgery (postoperative day [POD 1] 1) up through POD 3, unless discharge occurs first. The VR intervention will be offered to all participants at least once (for a maximum use of up to twice daily) up to six times. Each VR session will last up to no longer than 30 minutes. The length of each session will be dependent on the participant's selection of the virtual environment. Pain, anxiety, state of relaxation, and side effects will be measured before and after each VR session using pre-post questionnaires (Numeric rating scale for pain and relaxation and the Spielberger State Anxiety Inventory for anxiety). After each VR session, participants will be asked about side effects. All participants will be asked to complete the System Usability Scale (SUS) questionnaire before discharge. Additionally, a convenience sample of up to 15 patients from diverse groups will be asked about their experience with VR through a one-time one-on-one, 15-minute qualitative semi-structured interview & a user satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 65 years of age
2. expected to be hospitalized for at least 48 hours after an elective major surgery
3. able to speak, read, and understand English
4. following surgery, is deemed stable and recovered by post-anesthesia care unit (PACU) and admitted to a medical-surgical unit by at least postoperative day 2

Exclusion Criteria:

1. patients with severe/profound cognitive impairments (i.e., SPMSQ score of four or less)
2. patients with a history of self-reported motion sickness
3. current or prior diagnosis of epilepsy
4. injury or surgery to the eyes, face, or neck that prevents using a VR HMD
5. non-elective surgery (urgent or emergency surgery)
6. blindness or severe visual impairment
7. severe hearing loss
8. the VR system deemed inappropriate by the treating clinician
9. patient reports nausea, vomiting, or dizziness just prior to the VR session
10. acute illness preventing the use of the VR after surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Mean change from self-reported baseline pain immediately before using virtual reality on the 11-point Numeric Rating Scale (NRS) to immediately after using virtual reality | Pre/post virtual reality from 1-day post-surgery up to approximately 3 days post-surgery during hospitalization.
  The NRS is a validated unidimensional measure of self-reported pain intensity in adults after surgery. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing extreme pain. A change = pain score immediately after use of virtual reality - baseline pain score taken immediately prior to use of virtual reality. Self-reported pain scores using the NRS will be measured pre/post each time virtual reality is used, starting as early as 1-day following surgery up to approximately 3 days after surgery.

SECONDARY OUTCOMES:
Mean change from self-reported baseline state of relaxation immediately before using virtual reality on the 11-point Numeric Rating Scale (NRS) to immediately after using virtual reality | Pre/post virtual reality from 1-day post-surgery up to approximately 3 days post-surgery during hospitalization.
  The 11-point numeric scale ranges from '0' representing "Not relaxed at all" to '10' representing " As relaxed as one could imagine." A change = relaxation score using NRS immediately after use of virtual reality - baseline NRS relaxation score taken immediately prior to use of virtual reality. Self-reported relaxation scores using the NRS will be measured pre/post each time virtual reality is used, starting as early as 1-day following surgery up to approximately 3 days after surgery.
Mean change from self-reported baseline anxiety immediately before using virtual reality on the Spielberger State-Trait Anxiety Inventory (STAI) 5-item (STAI-5) to immediately after using virtual reality | Pre/post virtual reality from 1-day post-surgery up to approximately 3 days post-surgery during hospitalization.
  Each item on the STAI-5 is scored on a scale of 1 to 4 with 1 representing " Not al all," 2 representing "somewhat," 3 representing "moderately so," and 4 representing "very much so." A higher score indicates a higher level of anxiety. A change = total STAI-5 score immediately after use of virtual reality - baseline STAI-5 score taken immediately prior to use of virtual reality. Self-reported anxiety scores using STAI-5 will be measured pre/post each time virtual reality is used, starting as early as 1-day following surgery up to approximately 3 days after surgery.
Detection of virtual reality side effects immediately after using virtual reality | post virtual reality from 1-day post-surgery up to approximately 3 days post-surgery during hospitalization.
  A 5-item question survey with "yes" or "no" as response options, will be administered after each virtual reality session to determine participant self-reported side effects.
Determine self-reported usability of virtual reality using the System Usability Scale(SUS). | System Usability will be measured at one timepoint- from post-surgery day 1 to day 3.
  The System Usability Scale(SUS) is reliable tool for measuring usability. It consists of a 10-item questionnaire with five response options for respondents, with 1 representing "Strongly disagree" and 5 representing "Strongly agree". The participant's scores for each question are converted to a new number, added together, and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. A higher score indicates greater self-reported usability.
Determine the overall user experience with virtual reality as an adjunct for postoperative pain 1-3 days after surgery during hospitalization. | System Usability will be measured at one timepoint- from post-surgery day 1 to day 3.
  Using 8 questions as part of a semi-structured interview guide, the overall user experience with virtual reality will be described through inductive qualitative thematic analysis. A one-time 15-minute recorded one-to-one interview will occur at study completion. Questions are focused on understanding the overall user experience.
Determine user satisfaction with virtual reality using an 8-item survey. | User satisfaction with virtual realiuty will be measured at one timepoint- from post-surgery day 1 to day 3.
  Self-reported satisfaction scores (1 to 5; 1-totally disagree, 5-totally agree). A higher overall score indicates higher user satisfaction. The survey will be administered once at study completion prior to discharge.
Percentage of participants who complete all study questionnaires. | Completion of all study questionnaires will be measured at one time point- from study enrollment up until post-surgery 3 days.
  Compliance with questionnaire completion as measured by the proportion of recruited participants who use virtual reality at least once during the first 1-3 days post-surgery and complete all study questionnaires.
Percentage of older adults who declined to participate in the study. | Pre-intervention
  Of the total number of older adults recruited for the study, the percentage of those declining to participate will be recorded, along with the reason(s) for non participation in the study.
The percentage of virtual reality sessions started compared to the number of sessions offered. | Post-surgery day 1 to 3
  Determine the overall percentage of virtual reality sessions completed compared to the number of sessions offered. Each participant will be offered a virtual reality session up to twice daily post-surgery day 1 to 3 for a total of 6 sessions.
Duration of use for each virtual reality session | Post-surgery day 1 to 3
  Determine the mean duration of use.
Assessment of the ability to retain enrolled participants. | from 1-day post-surgery up to approximately 3 days post-surgery during hospita
  The proportion of enrolled participants who complete baseline questionnaires but do not start the first virtual reality session during 1-3 post-surgery.
Rate of discontinued interventions | Post-surgery day 1 to 3
  Determine the number of enrolled participants who do not complete more than one virtual reality session and the reason for discontinuing study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Park, PhD, NP, RN, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No